CLINICAL TRIAL: NCT02145624
Title: A Randomised Controlled Trial Comparing Two Pertussis-containing Vaccines in Pregnancy and Vaccine Responses in UK Mothers and Their Infants
Brief Title: A Trial Comparing Two Pertussis-containing Vaccines in Pregnancy and Vaccine Responses in UK Mothers and Their Infants
Acronym: iMAP2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health England (Other Government)
Collaborators: Institute of Child Health (Other); St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: iMAP2
Record Dates: First submitted 2014-05-13; First posted 2014-05-23 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2018-08

CONDITIONS: Responses to Infant Immunisations
Keywords: pertussis; maternal vaccination; maternal immunisation; immune response
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Repevax (Active Comparator): Repevax in pregnancy
  Interventions: Drug: Repevax
- Boostrix-IPV (Active Comparator): Boostrix-IPV in pregnancy
  Interventions: Drug: Boostrix-IPV
- unvaccinated (No Intervention): unvaccinated mothers

INTERVENTIONS:
Drug: Repevax — vaccine
  Other Names: Pertussis containing vaccine
  Arms: Repevax
Drug: Boostrix-IPV — vaccine
  Other Names: Pertussis containing vaccine
  Arms: Boostrix-IPV

SUMMARY:
Due to an unexpectedly high number of infant deaths from whooping cough in 2012, the Department of Health acted to protect newborns between birth and completion of primary immunisations, the period with greatest risk of disease.

Vaccination of pregnant women with whooping cough vaccine in the third trimester of pregnancy was instigated nationally, so that antibodies produced by the Mum would cross the placenta to the unborn child, giving them passive protection at the most vulnerable time. This antibody transfer has been known for some time but has not been compared between the two whooping cough vaccines being used in pregnancy. Any effect the raised antibody might have on infant responses to the vaccines given in the first few months of life has also not been measured. This is particularly important as the infant immunisations include some of the same components as the whooping cough vaccines, which include diphtheria, tetanus and polio. Previous studies have shown that high levels of antibody prior to vaccination may affect subsequent antibody responses. It is therefore important to assess whether administration of the whooping cough vaccine in pregnancy adversely affects the protection afforded by the infant vaccines, particularly to those which are similar, namely tetanus and diphtheria as well as meningitis C and Hib vaccines which include diptheria and tetanus components in their structures. This study will assess immune responses of mothers and their babies (~200 pairs) to their vaccinations and will allow the comparison of two whooping cough vaccines being used in pregnancy. This will be done by taking small amounts of blood, which is the only way to measure antibody levels (the proxy of the immune response), before and after the vaccinations. A group of unvaccinated women and their babies (50 pairs) will also be recruited to allow comparison of their immune responses.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women who, at the time of enrolment

• are aged 1645 years Infants of the women recruited will also be seen during the study. They will be given their immunisations according to the routine childhood immunisation schedule and will have blood samples collected as detailed in the clinical procedures section of this form. Their inclusion/ exclusion will be as per the Green Book recommendations by the UK Dept of Health.

Exclusion Criteria:

Participants may not be included in the study if any of the following apply:

All women:

* Bleeding disorder
* Receipt of any pertussis containing vaccine in the previous 12 months

Women to be vaccinated only (i.e. not the control group):

* Received immunoglobulin or other blood product within the preceding 3 months
* Fulfil any of the contraindications to vaccination specified in The Green Book on Immunisation (https://www.gov.uk/government/organisations/publichealthenglan d/series/immunisationagainstinfectiousdiseasethegreenbook), including:

  * A confirmed anaphylactic reaction to a previous dose of diphtheria, tetanus, pertussis or poliomyelitis containing vaccine
  * A confirmed anaphylactic reaction to any component of the vaccine
  * A confirmed anaphylactic reaction to a previous dose of diphtheria, tetanus, pertussis or poliomyelitis containing vaccine
  * Temporary Exclusion Criteria If the pregnant woman or the baby has an axillary/aural temperature ≥ 38°C, then vaccination and blood sampling will be postponed until resolution of fever. If the pregnant woman or baby is acutely unwell, vaccination will postponed until resolution. Blood sampling will also be postponed for seven days after completion of any antibiotic course.

Infants will be vaccinated under the routine national immunisation schedule in accordance with the inclusion/ exclusion criteria set out in the Department of Health "Green Book"

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 366 (Actual)
Dates: Start 2014-10; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
PT immunogenicity (IgG GMC) | Birth, 2, 5 and 13 months of age
  To compare antiPertussis Toxin (PT) IgG responses following primary immunisation with an acellular pertussiscontaining vaccine in infants born to mothers who received REPEVAX in pregnancy compared to infants whose mothers received BOOSTRIXIPV in pregnancy.
Immunogenicity of pertussis antigens (IgG GMC) | Birth, 2, 5 and 13 months of age
  To compare antibody responses to pertussis antigens (concentration of IgG antibody to PT, pertactin (PRN), filamentous haemagglutinnin (FHA) and fimbrial antigens 2 and 3 (FIM 2 and 3]), tetanus toxoid and diphtheria toxoid at birth amongst infants born to mothers who received REPEVAX in pregnancy compared to infants whose mothers received BOOSTRIXIPV in pregnancy
Immunogenicity of infant immunisations - pertussis antigens, meningococcal serogroup C, pnuemococcal vaccines at 2, 5 and 13 months of age, (all IgG GMC and SBA GMT for MenC) | Birth, 2, 5 and 13 months of age
  To compare antibody responses to pertussis antigens [IgG to PT, PRN, FHA and FIM 2 and 3], Hib antigen [PRP], tetanus toxoid and diphtheria toxoid; meningococcal serogroup C serum bactericidal antibody titres and meningococcal serogroup Cspecific IgG concentrations; 13 serotypespecific pneumococcal IgG concentrations and functional pneumococcal antibody studies at 2, 5 and 13 months of age (just before and one month after primary immunization and one month after booster vaccines) in infants born to mothers who received REPEVAX in pregnancy compared to infants whose mothers received BOOSTRIXIPV in pregnancy and compared to infants whose mothers who did not receive pertussis vaccination in pregnancy

OTHER OUTCOMES:
immunogenicity of pnuemococcal conjugate vaccine | birth, 2, 5 13 months
  immunogenicity of pnuemococcal conjugate vaccine
immunogenicity of meningococcal conjugate vaccine | birth, 2, 5, 13 months
  immunogenicity of meningococcal conjugate vaccine
immunogenicity of diphtheria vaccine | borth 2, 5, 13 months
  immunogenicity of diphtheria vaccine
immunogenicity of pertussis vaccination | birth, 2, 5, 13 months
  immunogenicity of pertussis vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Coates, PhD, Study Chair — Public Health England
Locations (3):
- United Kingdom (3):
  - Gloucestershire, Gloucestershire, Gloucestershire
  - Hertfordshire, Hertfordshire, Hertfordshire
  - St George's Vaccine Institute, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grassly NC, Andrews N, Cooper G, Stephens L, Waight P, Jones CE, Heath PT, Calvert A, Southern J, Martin J, Miller E. Effect of maternal immunisation with multivalent vaccines containing inactivated poliovirus vaccine (IPV) on infant IPV immune response: A phase 4, multi-centre randomised trial. Vaccine. 2023 Feb 10;41(7):1299-1302. doi: 10.1016/j.vaccine.2023.01.035. Epub 2023 Jan 21. PMID 36690561
- [Derived] Jones CE, Calvert A, Southern J, Matheson M, Andrews N, Khalil A, Cuthbertson H, Hallis B, England A, Heath PT, Miller E. A phase IV, multi-centre, randomized clinical trial comparing two pertussis-containing vaccines in pregnant women in England and vaccine responses in their infants. BMC Med. 2021 Jun 8;19(1):138. doi: 10.1186/s12916-021-02005-5. PMID 34098951
- See also: PHE website — https://www.gov.uk/government/organisations/public-health-england